CLINICAL TRIAL: NCT01667211
Title: A Single Center, Non-randomized, Open Phase II Clinical Study of Albumin-bound Paclitaxel Plus Nedaplatin in Patients With Advanced, Recurrent Metastatic Cervical Cancer
Brief Title: Clinical Study of Albumin-bound Paclitaxel Plus Nedaplatin in Cervical Cancer
Acronym: CSAPPPCC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Zhang rong, Chief Physician, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CH-GYN-001; 11-92/527 (Other: Cancer Institute and Hospital, CAMS)
Record Dates: First submitted 2012-07-10; First posted 2012-08-17 (Estimated); Last update posted 2012-08-22 (Estimated); Status verified 2012-08

CONDITIONS: Uterine Cervical Cancer
Keywords: Advanced uterine cervical cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Albumin-Bound Paclitaxel; nedaplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- albumin-bound paclitaxel plus nedaplatin (Experimental): albumin-bound paclitaxel plus nedaplatin: Intravenous albumin-bound paclitaxel, 175-200 mg/m2, d 1, was given every 3 weeks, combined with intravenous nedaplatin, 80- 100 mg/m2, d 2. At least 2 cycles will be completed for each patient, for whom responds to study treatment, 4-6 cycles will be completed.
  Interventions: Drug: albumin-bound paclitaxel plus nedaplatin

INTERVENTIONS:
Drug: albumin-bound paclitaxel plus nedaplatin — intravenous albumin-bound paclitaxel, 175-200 mg/m2, d 1, was given every 3 weeks, combined with intravenous nedaplatin, 80- 100 mg/m2, d 2. At least 2 cycles will be completed for each patient, for whom responds to study treatment, 4-6 cycles will be completed.
  Other Names: Abraxane (albumin-bound paclitaxel)

SUMMARY:
Using albumin-bound paclitaxel and nedaplatin in the advanced or recurrent metastasis cervical cancer, to evaluate the efficacy and toxic reaction.

DETAILED DESCRIPTION:
Albumin-bound paclitaxel is a novel, solvent-free, albumin-bound nanoparticle form of paclitaxel designed to avoid problems associated with solvents used in Taxol. And albumin-bound paclitaxel was characterized with high tolerated doses with greater efficacy, and with greater concentration in tumor tissue compared with normal tissues. This is a single center, non-randomized, open-label Phase II clinical study to investigate the efficacy and tolerability of albumin-bound paclitaxel plus nedaplatin in patients with advanced, recurrent metastatic cervical cancer. About 30 patients will receive 175-200 mg/m2 albumin-bound paclitaxel, d 1 combined with 80- 100 mg/m2 nedaplatin, d 2, every 3 weeks. At least 2 cycles will be completed for each patient, for whom responded to the treatment, 4-6 cycles will be completed.

ELIGIBILITY:
Inclusion Criteria:

* Cervical cancer, advanced or recurrent metastasis
* Measurable and assessible tumor lesions
* Used ordinary paclitaxel or platinum drugs, more than 28 days
* Aged 18-70
* KPS score> 60 points, expected to survive more than 3 months
* Normal bone marrow function
* The function of liver and kidney had no obvious damage
* Normal function of vital organs
* No brain metastases
* Patients or their agents to sign informed consent
* Compliance, and can be followed up regularly

Exclusion Criteria:

* Brain metastases
* Serious complications
* Acute inflammatory response
* Combined with other tumor
* Pregnancy or breast-feeding women
* Vertebral metastasis with nerve compression symptoms
* Large volume of pleural effusion, pericardial effusion
* Other malignancy within five years
* Drug allergy
* Other chemotherapy contraindications
* The possibility of pregnancy, and not willing to contraception
* No measurement of lesion
* Mental illness which is difficult to control

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2011-11; Primary Completion 2014-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
response rate | one year
  Percentage of patients who achieve partial response (PR)/ complete response (CR) based on RECIST

SECONDARY OUTCOMES:
Time to progression (TTP) | 2 years
  Measure of time from study treatment to disease progression
2-year progression-free survival (PFS) | 2 years
  Percentage of patients who have PFS two years after receiving study treatment.
safety and tolerability | 2 years
  Percentage of patients who experience an adverse event during this study.
Overall survival (OS) | 5 years
  Measure of time from study treatment to patient's death or lost to follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Rong Zhang, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Chinese Academy of Medical Sciences, Cancer Hospital, Gynecologic Oncology, Beijing, China